CLINICAL TRIAL: NCT04166968
Title: Multicenter Study on the Efficacy of Transcranial Direct Current Stimulation (tDCS) in Post-stroke Motor Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Collaborators: San Gerardo Hospital (Other); Maggiore Bellaria Hospital, Bologna (Other); Azienda Ospedaliero, Universitaria Pisana (Other); Fondazione Don Carlo Gnocchi Onlus (Other); Azienda Ospedaliera Universitaria Integrata Verona (Other); Azienda Unita Sanitaria Locale di Piacenza (Other); Azienda Ospedaliero Universitaria di Cagliari (Other); Ospedale Policlinico San Martino (Other); I.R.C.C.S. Fondazione Santa Lucia (Other); Catholic University of the Sacred Heart (Other); Istituti Clinici Zucchi (Other); Ospedali Riuniti di Foggia (Other)
Responsible Party: Principal Investigator, Carlo Miniussi, Professor, PhD, IRCCS Centro San Giovanni di Dio Fatebenefratelli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITSTUDYTDCS-45-2019
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Stroke, Ischemic; Stroke Hemorrhagic
Keywords: transcranial direct current stimulation; stroke rehabilitation
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The present study will be conducted in over 15 recruiting centers with a randomized double-blind design. Post-stroke patients will be randomly assigned to 3 parallel groups: Control Group (neuromotor training and sham stimulation), Experimental Group 1 (neuromotor training and cathodal tDCS over the unaffected hemisphere), Group 2 (neuromotor training and anodal tDCS over the affected hemisphere). Participants will be further partitioned on the basis of the acute/subacute and subacute/chronic stages (7-90 and 91 days from lesion onset, respectively).
Who Masked: Participant, Outcomes Assessor
Masking Description: Both participants and experimenters will be prevented from having knowledge of the assigned stimulation protocol. To do so, the investigator will create a series of numbers paired with real and sham interventions while the outcome assessor will be aware of the patient-number association only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Sham Comparator): neuromotor training and placebo stimulation
  Interventions: Device: Sham stimulation (sham-tDCS); Behavioral: Neuromotor training
- Group 1 (Experimental): neuromotor training and cathodal stimulation over the unaffected hemisphere
  Interventions: Device: Cathodal transcranial direct current stimulation (C-tDCS); Behavioral: Neuromotor training
- Group 2 (Experimental): neuromotor training and anodal stimulation over the affected hemisphere
  Interventions: Device: Anodal transcranial direct current stimulation (A-tDCS); Behavioral: Neuromotor training

INTERVENTIONS:
Device: Anodal transcranial direct current stimulation (A-tDCS) — Anodal tDCS will be performed for 20 minutes over the affected hemisphere with an intensity set to 2 mA
  Arms: Group 2
Device: Cathodal transcranial direct current stimulation (C-tDCS) — Cathodal tDCS will be performed for 20 minutes over the unaffected hemisphere with an intensity set to 2 mA
  Arms: Group 1
Device: Sham stimulation (sham-tDCS) — placebo stimulation
  Arms: Control Group
Behavioral: Neuromotor training — conventional neuromotor treatment

SUMMARY:
Several previous studies have used tDCS as a neuromodulation tool, showing improvements in several diseases (Lefaucheur et al., 2017). Based on these observations, it is believed that the use of tDCS in combination with specific motor training may provide the opportunity to induce behavioral improvements in patients with motor deficits. As shown in previous reports brain stimulation can, in fact, interact with the intrinsic ability of the brain to "repair" damaged brain functions, increasing the involvement of compensatory functional networks and thus inducing neuroplasticity. If these low-cost, easy-to-use stimulation techniques prove to be useful in improving motor deficits with long-term effects, the current study would open up new and interesting avenues in the field of neurorehabilitation. Given the potential long-lasting effects of tDCS, there is currently a growing interest in the clinical sector with the aim to reduce motor deficits in patients with brain injury. The most widely used protocols in stroke patients include the application of either anodal on the hypsilesional hemisphere or cathodal tDCS on the unaffected hemisphere (contralateral), so as to increase and decrease the excitability of the motor cortex, respectively (Nitsche and Paulus, 2001).

The main objective of this study is to evaluate the effectiveness of transcranial direct current stimulation in enhancing the functional recovery of the upper limb of stroke patients after three weeks of neuromotor training and subsequent follow-up. The secondary objective is to evaluate the treatment effects on balance, gait, motor dexterity and disability, besides the functional recovery of the lower limb.

ELIGIBILITY:
Inclusion Criteria:

* First-ever ischemic stroke
* Red or white stroke
* Barthel Index > 90 before lesion onset

Exclusion Criteria:

* Previous inborn neurological disease
* Previous acquired neurological disease
* Previous or current major psychiatric illness
* Epilepsy or anticonvulsant treatment
* Use of calcium channel blocker drugs
* Treatments with other technologies (robotics, FES, etc.)
* Neurolytic treatments with botulinum toxin

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline Fugl Meyer Assessment Scale (FMA) | End of 1st week; End of 2nd week; End of 3rd week; 90 days follow-up
  Performance-based assessment of sensorimotor impairment

SECONDARY OUTCOMES:
Changes from Baseline Box & Block Test (B&B) | End of 1st week; End of 2nd week; End of 3rd week; 90 days follow-up
  test for manual dexterity of upper extremity function
Changes from Baseline Barthel Index (BI) | End of 1st week; End of 2nd week; End of 3rd week; 90 days follow-up
  measure of daily living activities in relation to personal care and mobility of the patient
Changes from Baseline Trunk Control Test (TCT) | End of 1st week; End of 2nd week; End of 3rd week; 90 days follow-up
  assessment of the deteriorations in trunk control
Changes from Baseline Berg Balance Scale ( BBS) | End of 1st week; End of 2nd week; End of 3rd week; 90 days follow-up
  test of a person's static and dynamic balance abilities
Changes from Baseline 10 Meters Walking Test | End of 1st week; End of 2nd week; End of 3rd week; 90 days follow-up
  evaluation of functional mobility, gait, and vestibular function
Changes from Baseline Functional Ambulatory Classification (FAC) | End of 1st week; End of 2nd week; End of 3rd week; 90 days follow-up
  clinically meaningful outcome measure of mobility

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Miniussi, PhD, Principal Investigator — IRCCS Centro San Giovanni di Dio Fatebenefratelli
Locations (1):
- IRCCS Centro San Giovanni di Dio Fatebenefratelli, Brescia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided